CLINICAL TRIAL: NCT00046670
Title: Sleep Disordered Breathing, APOE, and Lipid Metabolism
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1191; R01HL071515 (NIH)
Record Dates: First submitted 2002-09-30; First posted 2002-10-01 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-03

CONDITIONS: Sleep Apnea Syndromes; Lung Diseases
MeSH Terms: conditions — Sleep Apnea Syndromes; Lung Diseases

SUMMARY:
To examine the relationship between obstructive sleep apnea and lipid metabolism.

DETAILED DESCRIPTION:
BACKGROUND:

Recent findings suggest interrelationships between obstructive sleep apnea, lipid metabolism, and neurodegeneration. Apolipoprotein E epsilon4 (APOE e4), a genetic marker linked to increased cardiovascular disease (CVD) risk and Alzheimer's disease (AD), is associated with a two fold increased risk of sleep disordered breathing (SDB), and an increase in severity of apnea symptoms. Preliminary data suggest that this association is stronger between the ages of 50 and 65. Other experiments suggest dysregulated leptin levels in obstructive sleep apnea (OSA). Taken together, these findings suggest common pathophysiological mechanisms involving dysregulated lipid metabolism in OSA. An understanding of these mechanisms is essential for the prevention and treatment of SDB.

DESIGN NARRATIVE:

Using case/control and family designs, the study: 1) extends the finding that apolipoprotein E epsilon4 (APOE e4) increases the risk of sleep apnea in the general population; 2) examines if polymorphisms in other genes regulating lipid levels are associated with sleep apnea; 3) studies the relationship between lipid regulatory gene polymorphisms, lipid profile (LDL- cholesterol, HDL-cholesterol, triglycerides), plasma leptin (and other lipid regulatory hormones), and sleep apnea levels.

T

ELIGIBILITY:
No eligibility criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2002-09; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Mignot — Stanford University

REFERENCES:
- [Background] Lin L, Finn L, Zhang J, Young T, Mignot E. Angiotensin-converting enzyme, sleep-disordered breathing, and hypertension. Am J Respir Crit Care Med. 2004 Dec 15;170(12):1349-53. doi: 10.1164/rccm.200405-616OC. Epub 2004 Sep 24. PMID 15447944
- [Background] Gottlieb DJ, DeStefano AL, Foley DJ, Mignot E, Redline S, Givelber RJ, Young T. APOE epsilon4 is associated with obstructive sleep apnea/hypopnea: the Sleep Heart Health Study. Neurology. 2004 Aug 24;63(4):664-8. doi: 10.1212/01.wnl.0000134671.99649.32. PMID 15326239
- [Background] Taheri S, Lin L, Austin D, Young T, Mignot E. Short sleep duration is associated with reduced leptin, elevated ghrelin, and increased body mass index. PLoS Med. 2004 Dec;1(3):e62. doi: 10.1371/journal.pmed.0010062. Epub 2004 Dec 7. PMID 15602591